CLINICAL TRIAL: NCT01432704
Title: Phase IV Study of Colecalciferol as an Add-on Treatment to Subcutaneously Administered Interferon-beta-1b for Treatment of MS
Brief Title: Colecalciferol as an Add-on Treatment to Subcutaneously-Administered Interferon-beta-1b for Treatment of Multiple Sclerosis (MS)
Acronym: 100207MS-H
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Merja Soilu-Hänninen, MD, PhD, neurologist, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2007-001958-99
Record Dates: First submitted 2011-08-16; First posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Sclerosis
Keywords: MS; vitamin D; environment
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- placebo capsules (Placebo Comparator): Identically appearing placebo capsules not containing colecalciferol
  Interventions: Drug: colecalciferol
- colecalciferol capsules (Active Comparator): Once weekly peroral colecalciferol capsules (Dekristol®, Swiss-Caps, Switzerland) containing 20 mg of colecalciferol corresponding to 20000 IU or 0.5 mg of vitamin D3 for a duration of 12 months
  Interventions: Drug: colecalciferol

INTERVENTIONS:
Drug: colecalciferol — Once weekly peroral colecalciferol capsules (Dekristol®, Swiss-Caps, Switzerland) that contain 20 mg of colecalciferol corresponding to 20000 IU or 0.5 mg of vitamin D3 for a duration of 12 months
  Other Names: (Dekristol®, Swiss-Caps, Switzerland)

SUMMARY:
This is a one-year multi-centre, double blind, placebo controlled, randomized trial investigating oral vitamin D3 (Colecalciferol) as an add-on treatment to interferon-beta-1b for Multiple Sclerosis (MS). Not less than one month after initiation of therapy with interferon beta 1b, MS patients will be randomised to once weekly treatment with peroral colecalciferol capsules (Dekristol®, Swiss-Caps, Switzerland) containing 0.5 mg of vitamin D3, or to once weekly peroral treatment with matching placebo. The hypothesis is that vitamin D suppresses clinical and MRI activity of MS.

DETAILED DESCRIPTION:
The patients will be examined clinically at baseline and at 6, and 12 months. Laboratory assessments will be performed at screening and 1, 2, 3, 6, 9 and 12 months after baseline. MRI will be performed (T1-weighted and T2-weighted) at randomization and 12 months thereafter. Sample size is 80 patients: two groups with 40 patients in each group. The primary statistical analyses will be based on the intent-to-treat (ITT) population which consist of all randomized patients who have started study medication. The primary efficacy variable MRI T2 BOD will be analyzed using ANCOVA with MRI T2 BOD at baseline as covariate. The incidence (with corresponding 95% confidence interval) of hypercalcaemia (mild, moderate and severe), laboratory abnormalities, dose adjustments, and significant adverse events will be calculated. The vitamin D status (proportion of patients with P-PTH <20 ng/l and S-OH(D)2 >85 nmol/l) at 6 and 12 months will be analyzed using logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* RRMS EDSS 0-5
* Betaferon used for at lest one month with positive MxA-response

Exclusion Criteria:

* hypercalcaemia
* kidney stones
* uncontrolled hypertension
* hypothyreosis
* peanut allergy
* severe depression
* sarcoidosis
* use of other IMD than interferon-beta

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of add-on -treatment with colecalciferol of MS patients treated with interferon beta-1b and | one year
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability
To estimate the effect of interferon-beta-1b with an add-on of colecalciferol versus interferon-beta-1b with an add-on of placebo on MRI T2 BOD at 12 months in comparison with MRI T2 BOD at baseline | 12 months

SECONDARY OUTCOMES:
Number of Gadolinium-enhancing lesions on T1 and /or new enlarging lesions on T2/PD based on MRI done 12 months following randomisation compared with the MRI done at the time of randomisation | 12 Months